CLINICAL TRIAL: NCT04870164
Title: A Phase 1, First-time-in-human, Dose Ascending Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MP0420 (a Novel Drug Candidate With Potential for Treatment of COVID-19) in Healthy Volunteers
Brief Title: Safety, Tolerability and PK of Ensovibep (MP0420 - a New Candidate With Potential for Treatment of COVID-19)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to hypersensitivity observed in 3 subjects, although no stopping rules were met, the Sponsor decided to halt recruitment for further investigation. After analysis of PK, i.m. administration was not required, and recruitment stopped.
Sponsor: Molecular Partners AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: MP0420-CP101; 2020-004365-39 (EudraCT Number)
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: ensovibep; COVID-19 treatment; SARS-CoV-2; Corona; designed ankyrin repeat protein (DARPin®); angiotensin-converting enzyme 2 (ACE2)
MeSH Terms: conditions — COVID-19 | interventions — ensovibep; Designed Ankyrin Repeat Proteins; COVID-19 Drug Treatment

STUDY DESIGN:
Intervention Model Description: Parallel (Part A) Sequential (Part B and Part C)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A only
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- ensovibep dose 1 (infusion) (Experimental)
  Interventions: Drug: Ensovibep
- ensovibep dose 2 (infusion) (Experimental)
  Interventions: Drug: Ensovibep
- ensovibep dose 3 (infusion) (Experimental)
  Interventions: Drug: Ensovibep
- placebo (infusion) (Placebo Comparator)
  Interventions: Drug: Placebo
- ensovibep dose 4 (IV bolus) (Experimental)
  Interventions: Drug: Ensovibep
- ensovibep dose 5 (IV bolus) (Experimental)
  Interventions: Drug: Ensovibep
- ensovibep dose 6 (SC injection) (Experimental)
  Interventions: Drug: Ensovibep
- ensovibep dose 7 (SC injection) (Experimental)
  Interventions: Drug: Ensovibep
- ensovibep dose 8 (SC injection) (Experimental)
  Interventions: Drug: Ensovibep
- ensovibep dose 9 (SC injection) (Experimental)
  Interventions: Drug: Ensovibep
- ensovibep dose 10 (IM injection) (Experimental)
  Interventions: Drug: Ensovibep
- ensovibep dose 11 (IM injection) (Experimental)
  Interventions: Drug: Ensovibep
- ensovibep dose 12 (IM injection) (Experimental)
  Interventions: Drug: Ensovibep
- ensovibep dose 13 (IM injection) (Experimental)
  Interventions: Drug: Ensovibep

INTERVENTIONS:
Drug: Ensovibep — The study will start with a low-dose cohort and after a safety review escalate to the higher dose cohorts. 3 IV infusion, 2 IV bolus, 4 subcutaneous and 4 intramuscular cohorts are planned. Subjects receive one or two administration(s) on day 1, depending on the cohort.
  Other Names: MP0420; DARPin; COVID-19 treatment
  Arms: ensovibep dose 1 (infusion); ensovibep dose 10 (IM injection); ensovibep dose 11 (IM injection); ensovibep dose 12 (IM injection); ensovibep dose 13 (IM injection); ensovibep dose 2 (infusion); ensovibep dose 3 (infusion); ensovibep dose 4 (IV bolus); ensovibep dose 5 (IV bolus); ensovibep dose 6 (SC injection); ensovibep dose 7 (SC injection); ensovibep dose 8 (SC injection); ensovibep dose 9 (SC injection)
Drug: Placebo — One administration at day 1 by infusion.
  Arms: placebo (infusion)

SUMMARY:
This study will investigate how ensovibep is distributed throughout the body, the safety and the tolerability of ensovibep in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between ages of 18-65 years
* Body mass index of 18.0-35.0 kg/m2
* Non-smokers for at least 3 months
* Deemed healthy on the basis of a clinical history, physical examination, ECG, vital signs, and laboratory tests of blood and urine
* Agree to follow the contraception requirements of the trial
* Able to give fully informed written consent.

Exclusion Criteria:

* Positive tests for hepatitis B & C, HIV
* Severe adverse reaction to any drug
* Drug or alcohol abuse
* Use of over-the-counter medication (with the exception of paracetamol [acetaminophen]) during the 7 days before the first dose of trial medication, or prescribed medication during the 28 days before first dose of trial medication
* Any vaccination within 4 weeks before dose of trial medication
* Participation in other clinical trials of unlicensed medicines within the previous 3 months
* Loss of more than 400 mL blood within the previous 3 months
* Vital signs outside the acceptable range
* Clinically relevant abnormal findings at the screening assessment
* Acute or chronic illness
* Clinically relevant abnormal medical history or concurrent medical condition
* Possibility that volunteer will not cooperate
* Females who are pregnant or lactating, or who are sexually active and not using a reliable method of contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Vital Signs: Blood Pressure Systolic and Diastolic (mmHg) | up to day 100 (EOS)
Vital Signs: Heart Rate (bmp) | up to day 100 (EOS)
Vital Signs: Tympanic Temperature (°C) | up to day 100 (EOS)
Vital Signs: Oxygen Saturation (SpO2%) | up to day 100 (EOS)
Cardiac Safety assessed by 12-lead Electrocardiogram (ECG) | up to day 100 (EOS)
Physical Examination | up to day 100 (EOS)
  For safety purpose, the following will be examined during full physical examinations: general appearance; head, ears, eyes, nose and throat; thyroid; lymph nodes; back and neck; heart; chest; lungs; abdomen; skin; and extremities; and the following systems will be assessed: musculoskeletal and neurological.
Number of subjects with Laboratory Abnormalities | up to day 100 (EOS)
Assessment of local tolerability | up to day 100 (EOS)
  Number of subjects with reaction at the injection site. The injection site is assessed for any pain, tenderness, erythema and induration.
Number of subjects with Adverse Events | up to day 100 (EOS)

SECONDARY OUTCOMES:
Observed maximum concentration (Cmax) | up to day 100 (EOS)
  The maximum observed concentration (Cmax) is estimated based on the serum concentrations.
Time to Cmax (Tmax) | up to day 100 (EOS)
The area under the serum concentration-time curve (AUC) | up to day 100 (EOS)
Apparent total body clearance of the drug from plasma (CL) | up to day 100 (EOS)
The apparent volume of distribution during terminal phase after drug administration (Vz) | up to day 100 (EOS)
Terminal Elimination Half-Life (T½) | up to day 100 (EOS)
Proportion of subjects with treatment-emergent anti-drug antibodies (ADA) | up to day 100 (EOS)

CONTACTS AND LOCATIONS:
Locations (1):
- HMR, London, United Kingdom